CLINICAL TRIAL: NCT06302439
Title: A Prospective Observational Patient Registry to Evaluate Disease Progression in Patients With ENPP1 Deficiency and Infantile-Onset ABCC6 Deficiency (GACI Type 2)
Brief Title: PROPEL - A Prospective Observational Patient Registry to Evaluate ENPP1 and ABCC6 Deficiency
Status: Recruiting | Type: Observational
Sponsor: Inozyme Pharma (Industry)
Collaborators: GACI Global (Unknown)
Responsible Party: Sponsor
Other Study IDs: INZ701-007
Record Dates: First submitted 2024-02-16; First posted 2024-03-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ectonucleotide Pyrophosphatase/Phosphodiesterase 1 Deficiency; ATP-Binding Cassette Subfamily C Member 6 Deficiency
Keywords: Ectonucleotide pyrophosphatase; ENPP1; Generalized Arterial Calcification of Infancy; GACI; Autosomal Recessive Hypophosphatemic Rickets Type 2; ARHR2; Observational; Registry; ATP-Binding Cassette Subfamily C Member 6 Deficiency; ABCC6; PROPEL; Phosphodiesterase 1
MeSH Terms: conditions — Arterial calcification of infancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention for this observational study — No Intervention for this observational study

SUMMARY:
The purpose of this prospective registry is to characterize the natural history of ectonucleotide pyrophosphatase/phosphodiesterase1(ENPP1) Deficiency and the infantile-onset form of adenosine triphosphate (ATP) binding cassette transporter protein subfamily C member 6 (ABCC6) Deficiency longitudinally. The registry will prospectively gather information about the genetic, biochemical, physiological, anatomic, radiographic, and functional manifestations (including patient reported outcomes [PROs]) of each disease during routine, standard-of-care visits, with the aim of developing a comprehensive understanding of the burden of illness and progressive nature of the disease.

DETAILED DESCRIPTION:
ENPP1 Deficiency is a rare, genetic disorder caused by inactivating mutations in the ENPP1 gene that encodes the ENPP1 enzyme. Infantile-onset ENPP1 Deficiency has a high mortality (approximately 50%) in the first 0 to 6 months of life, a result of downstream cardiopulmonary complications. Pediatric patients with ENPP1 Deficiency typically experience rickets, a condition also known as autosomal-recessive hypophosphatemic rickets type 2 (ARHR2), while adults experience osteomalacia (softened bones), and they can exhibit a range of signs and symptoms that include hearing loss, arterial calcification, and cardiac and/or neurological involvement.

Like ENPP1 Deficiency, infantile-onset ABCC6 Deficiency is a rare, genetic disorder caused by mutations in the ABCC6 gene. Infantile-onset of ABCC6 Deficiency resembles the acute infantile form of ENPP1 Deficiency. Pediatric patients with biallelic or monoallelic ABCC6 mutations can present with cerebrovascular disease.

This is an international, multicenter, prospective, non-interventional, observational registry of patients with biallelic variants in ENPP1, symptomatic patients with monoallelic ENPP1 variants and the infantile-onset form of ABCC6 Deficiency (<18 years of age). The registry will include patients with ENPP1 Deficiency or infantile-onset of ABCC6 Deficiency independent of treatment regimen. Note: patients participating in an INZ-701 interventional clinical study are not eligible.

Registry participation will consist of a Screening Period and an Observational Period. During the Screening Period, both retrospective data (past medical history) and data available at the time of consent (baseline visit) will be collected. Data collected will include standard of care assessments, which may consist of any or all of the following: laboratory testing, radiographical assessment of calcification and vascular stenosis, bone mineralization, with addition of performance outcomes, patient-, caregiver-, and physician-reported outcomes, and healthcare utilization. During the Observational Period, participants will be assessed during their routine visits for changes in their disease and PROs and data will be added periodically to the database. There will be an opportunity for an optional blood draw to assess levels of inorganic pyrophosphate (PPi) at each routine visit.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate must meet all the following inclusion criteria:

1. Must provide written or electronic consent after the nature of the registry has been explained, and prior to any research-related procedures, per International Council for Harmonisation (ICH) Good Clinical Practice (GCP)
2. Agree to provide access to relevant medical records
3. One of the following genetic or clinical criteria

   1. A confirmed prenatal or postnatal molecular genetic diagnosis of ENPP1 Deficiency with biallelic mutations (ie, homozygous or compound heterozygous) performed by a College of American Pathologists/Clinical Laboratory Improvement Amendments (CAP/CLIA) certified laboratory or regional equivalent

      OR
   2. Monoallelic ENPP1 mutation confirmed by a certified CAP/CLIA laboratory or regional equivalent and any of the following clinical symptoms:

   i. ≥ 1 traumatic vertebral fracture

ii. ≥ 2 fractures as an adult (eg, long-bones, digits, vertebrae)

iii. Low bone mineral density (dual-energy X-ray absorptiometry [DXA] Z-score <1.5) and <55 years of age

iv. Bone or joint pain interfering with movement or daily activities

v. History of myocardial infarction (MI), unstable angina, transient ischemic attack (TIA) or low cardiac output before the age of 40 yrs.

vi. History of rickets or bone deformity

vii. Diagnosis of ossification of the posterior longitudinal ligament (OPLL)

viii. Other clinical symptoms, with approval by Inozyme

OR

c. A confirmed prenatal or postnatal molecular genetic diagnosis of ABCC6 Deficiency with biallelic mutations confirmed by a certified CAP/CLIA laboratory or regional equivalent, and <18 years of age

Exclusion Criteria:

Individuals who meet the following exclusion criteria will not be eligible to participate:

1. Participant or their legally designated representative does not have the cognitive capacity to provide informed consent
2. Patients who are currently participating in an INZ-701 interventional clinical study, with the exception of expanded access programs and long-term safety follow-up studies

   1. Participants in interventional studies may be approached for inclusion in the registry once their involvement in the treatment period of the clinical study has been completed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Evidence of biallelic ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) variants in ENPP1 Deficiency
  or
  Evidence of monoallelic ENPP1 variants and disease-related symptoms
  or
  Infantile onset with biallelic adenosine triphosphate (ATP) binding cassette transporter protein subfamily C member 6 (ABCC6) variants in participants aged <18 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2034-05 (Estimated); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
Characterization of the natural history of ENPP1 Deficiency and the infantile-onset form of ABCC6 Deficiency longitudinally | Annually up to 10 years
  Assessments will be collected during each subject's routine visit. The assessments will be done per local standard of care.
Assessment of Patient Functional changes through a validated Patient Reported Outcomes (PROs) tool | Annually up to 10 years
  For each subject, patient function will be assessed using the appropriate Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaires. These may include: PROMIS Cognitive Function, PROMIS Fatigue, PROMIS Pain Intensity, PROMIS Pain Interference and PROMIS Physical Function. Each questionnaire is scored on a 5-point Likert scale ranging from 1 (never) to 5 (always). High scores indicate more of the domain being measured (eg, more fatigue, more physical function). Raw scores are converted to T-Scores based on a mean of 50 and a standard deviation of 10, allowing comparison of the sample to the general population.
  Parent Proxy questionnaires will be used for children aged 5 to <18 years
Assessment of Health-Related Quality-of-Life (HRQoL) changes through validated Patient Reported Outcomes (PROs) tools | Annually up to 10 years
  For each subject, HRQoL will be assessed using the following scales:
  age 5 to <18 years: Pediatric QoL scales (Short Form [SF]-10, Caregiver Global Impression of Status/Severity [CaGI-S]);
  age ≥18 years: Adult QoL scales (Short Form [SF]-36, Patient Global Impression of Status/Severity [PGI-S])
  The SF-10 is a 10-item caregiver-completed questionnaire for assessment of physical and psychosocial HRQoL in children. Each question has 5 options ranging from "Excellent" to "Poor". Higher scores are associated with better HRQoL.
  The SF-36 measures a broad spectrum of physical and mental health domains, including physical functioning, role limitations due to physical and emotional problems, bodily pain, general health perceptions, vitality, social functioning, and emotional well-being. The SF-36 generates scores ranging from 0-100 with higher scores associated with better HRQoL.
  The CaGI-S and PGI-S will be scored across a 7-point scale with lower scores associated with better HRQoL.
Measurement of inorganic phosphate (PPi) levels in patients' venous blood | Annually up to 10 years
  For each subject, QoL will be assessed using the following scales: global clinical impression of severity (GCI-S) and, short form 10 health survey for children and short form 36 health survey for adults short form 10 health survey for children and short form 36 health survey for adults

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - CLINILABS Drug Development Corp, Eatontown, New Jersey
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
- CHU Sainte-Justine Research Centre, Montreal, Quebec, Canada
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- IRCCS San Raffaele Hospital - Main, Milan, Italy
- The University of Tokyo Hospital, Tokyo, Japan
- Royal Hospital Muscat, Muscat, Oman
- Spain (2):
  - EU Hub - VCTC, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
- Umraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)
- VCTC, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided